CLINICAL TRIAL: NCT02687334
Title: Changes of Cerebral Oxygenation During Anesthesia Induction
Status: Completed | Type: Observational
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Associate proffesor, China Medical University, China
Other Study IDs: 2015110301
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-02

CONDITIONS: Cerebral Oxygen Saturation
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Standard general anesthesia induction: Patients scheduled for elective surgery at the First Hospital of China Medical University will be recruited for the study beginning in February 2016.We will investigate the changes of cerebral oxygenation during anesthesia induction of standard general anesthesia
  Interventions: Drug: 100% Oxygen

INTERVENTIONS:
Drug: 100% Oxygen — We will investigate the changes of cerebral oxygenation during anesthesia induction of standard general anesthesia with 100% oxygen

SUMMARY:
The aim of this study was to investigate the changes of cerebral oxygen saturation (rSO2) during anesthesia induction.

DETAILED DESCRIPTION:
The aim of this study was to investigate the relationship between the cerebral oxygen saturation (rSO2) and pressure of carbon dioxide (PaCO2) and oxygen (PaO2) in arterial blood and to identify the covariates between rSO2 and PaCO2 and PaO2 during the period of anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if they were ethnic Chinese, between 18 and 65 years old, American Society of Anesthesiologists (ASA) physical status I or II, and undergoing a radical operation for mastocarcinoma.

Exclusion Criteria:

* Patients were excluded if they had a body mass index exceeding 30 kg/m2, had a history of hypertension or diabetes mellitus, or were allergic to anesthesia drugs used in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients scheduled for elective radical operations for mastocarcinomaat in the First Hospital of China Medical University will be recruited for the study
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
changes of cerebral oxygen saturation | Baseline and 30 minutes
  the relationship between the cerebral oxygen saturation (rSO2) and pressure of carbon dioxide (PaCO2) and oxygen (PaO2) in arterial blood

CONTACTS AND LOCATIONS:
Overall Officials: Wen-fei Tan, M.D.,PhD., Principal Investigator — the First Hoapital of China Medical University
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes